CLINICAL TRIAL: NCT07338305
Title: The Copenhagen Translational Skin Immunology Biobank and Research Program - BIOSKIN: Methotrexat to Hand Eczema
Brief Title: Methotrexat to Hand Eczema in the BIOSKIN Cohort
Acronym: BIOSKIN: MTX
Status: Active, not recruiting | Type: Observational
Sponsor: Lone Skov (Other)
Collaborators: University of Copenhagen (Other); Herlev and Gentofte Hospital (Other)
Responsible Party: Sponsor-Investigator, Lone Skov, Professor, MD., Copenhagen University Hospital at Herlev
Organization: Copenhagen University Hospital at Herlev (Other)
Other Study IDs: H-21032986; LFST21500002 (Other Grant/Funding Number: The LEO fundation); No grant number (Other Grant/Funding Number: The Copenhagen University Hospital, Herlev and Gentofte Hospital, Denmark)
Record Dates: First submitted 2025-11-27; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis; Contact Dermatitis; Hand Eczema
Keywords: Skin immunology; Real-life
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis, Contact

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic hand eczema: Patients diagnosed with chronic hand eczema and initiating treatment with systemic methotrexat enrolled for longitudinal clinical biological follow-up in a real-life setting.

SUMMARY:
Handeczema is a common chronic skin disease that markedly affect health and quality of life. Effective treatment is limited by the lack of biomarkers that can predict disease course, comorbidities and treatment response. This study is is an observational, prospective, study of patients initiating treatment with methotrexat at the Department of Dermatology and Allergy at Herlev- and Gentofte Hospital.

The main aim is to study the clinical effect of methotrexat in patients with hand eczema. Secondary aims are to study drug survival, reasons for termination of treatment and side effects.

DETAILED DESCRIPTION:
The Copenhagen Translational Skin Immunology Biobank and Research Programme (BIOSKIN) is a prospective translational biobank and research study designed to recruit 3,000 patients with atopic dermatitis, allergic contact dermatitis or psoriasis over at least five years. The open longitudinal study design allows participants to enter and leave the cohort at time points that reflect their natural disease and treatment course. At each study visit, investigators collect biological samples, conduct structured interviews, and obtain patient-reported outcomes on disease-specific and general health-related factors.

In this study of patients initiating treatment with methotrexat because of hand eczema, patients are assessed with clinical assessments including dermatologist-verified diagnose, evaluation of disease severity, and detailed phenotyping. Examinations are performed before and after initiation of methotrexat as a tablet or as subcutaneous injections, and at least annually.

Longitudinal modelling will enable detailed characterisation of the patiens and disease trajectories and treatment responses. The aim is to improve understanding of the effect and sideeffects of methotrexat in a cohort of hand eczema patients with moderate to severe disease.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of any age with psoriasis, atopic dermatitis, contact dermatitis, or other inflammatory skin diseases.
* Patients seen at the Department of Dermatology and Allergy, Herlev and Gentofte Hospital, or recruited through public advertisement.
* Ability to provide informed consent (parent/guardian for minors).
* Healthy volunteers

Exclusion Criteria:

* Inability or unwillingness to provide informed consent.
* Any condition that, in the investigator's judgment, makes participation inappropriate or unsafe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Department of Dermatology and Allergy, Herlev and Gentofte Hospital,
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Longitudinal Clinical Disease Activity: Hand Eczema Severity Index (HECSI) | baseline to at least 5 years
  A validated clinical scoring system used to assess the severity and extent of hand eczema based on clinical signs and area involved, will be used

SECONDARY OUTCOMES:
Patient Reported Outcome: Dermatology Life Quality Index (DLQI) | Baseline to at least 5 years
  A validated patient-reported questionnaire measuring the impact of skin disease on quality of life.
Clinical characteristics | Baseline to at least 5 years
  Baseline characteristics of included patients for example if they are current smokers, if they have wet work, previous systemic treatments, registred etiology and morphology and duration of hand eczema and disease activity.
Allergic and genetic characteristics | At least 5 years
  Filaggrin mutation status, and positive patch/skin prick tests; and total serum IgE level from blood samples.
Drug survival and side effects | From baseline to at least 5 years
  Treatment duration, side effects and reasons for discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Lone Skov, Professor, Study Director — Department of Dermatology and Allergy, Herlev and Gentofte Hospital
Locations (1):
- Department of Dermatology and Allergy, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to restrictions under the Danish Data Protection Act and related regulations, which do not permit the disclosure of identifiable or potentially identifiable health data to external parties.

REFERENCES:
- [Background] Lovendorf MB, Johansen JD, Skov L. BIOSKIN: A Protocol for the Copenhagen Translational Skin Immunology Biobank and Research Programme. BMJ Open. 2024 Feb 24;14(2):e077207. doi: 10.1136/bmjopen-2023-077207. PMID 38401898
- See also: Website for participants, researchers and patients — https://www.bioskin.dk/